CLINICAL TRIAL: NCT06504173
Title: Use of Diced Cartilage for Management of Internal Mammary Vessel Exposure Sites in Autologous Breast Reconstruction
Brief Title: Diced Cartilage in Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: ISAR Klinikum (Other)
Collaborators: Breast Imaging Division, Radiologie Augsburg Friedberg / Breast Center Augsburg, Augsburg, Germany (Unknown)
Responsible Party: Principal Investigator, Peter Paul Pfeiler, MD, Consultant, ISAR Klinikum
Other Study IDs: DIC-RIP
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mammaplasty; Microsurgery; Rip Reconstruction Cartilage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diced cartilage (DC): After removing a part of the rip cartilage and microsurgery, the exposed internal mammary vessels in autologous free flap breast reconstruction was restored with diced cartilage (DC) out of the removed rip cartialge.
  Interventions: Procedure: diced cartilage
- control: After removing a part of the rip cartilage and microsurgery, the exposed internal mammary vessels in autologous free flap breast reconstruction was NOT restored.

INTERVENTIONS:
Procedure: diced cartilage — In reconstructions using DC management of IMVES, the surgical nurse processed the removed cartilage into DC using a dermatome blade. Cartilage pieces of approximately 0,5-1 mm were used. After microvascular anastomosis (coupler device for venous anastomosis; Synovis MCA, Birmingham AL, USA), all DC was placed back into the rib removal zone using a blunt dissector. The vessels were embedded and stabilized in cartilage paste according to the desired orientation.
  Groups: diced cartilage (DC)

SUMMARY:
Exposure of internal mammary vessels in autologous breast reconstruction often requires removal of a rib cartilage segment, which can lead to contour deformity in the craniomedial breast pole. This study evaluated the use of diced cartilage (DC) to counteract substance loss in the microvascular anastomosis area, and investigated safety and suitability of the procedure to avoid postoperative deformities.

DETAILED DESCRIPTION:
This retrospective, single-center cohort study included all breast reconstructions in which DC was used from October 2021 to June 2023. Reconstructions using DC were subdivided based on previous exposure to breast radiotherapy (DC vs. DCR). The control group consisted of an equal number of consecutive reconstructions performed prior to the use of DC. The effect of DC on breast contour preservation was investigated using breast magnetic resonance imaging (MRI; > 6 months post-op) and photographic documentation (6-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Autologous free flap breast reconstruction using the internal mammary vessels as recipient vessels from October 2021 to June 2023
* MRI subcohort: Magnetic resonance imaging (MRI) scans performed at least 6 months postoperatively

Exclusion Criteria:

* Autologous free flap breast reconstruction using a perforator of the internal mammary vessels as recipient vessels from October 2021 to June 2023
* Autologous free flap breast reconstruction using the thoracodorsal vessels as recipient vessels from October 2021 to June 2023

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The limitation of this study to the female gender is due to the phenotypic anatomical body structure and the intended reconstruction.
Study Population: The study population consists of women who received autologous free flap breast reconstruction using internal mammary vessels as recipient vessels.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance imaging (MRI) scans: soft tissue sinking of the recipient vessels area | October 2021 to June 2023
  the sinking depth of epicostal soft tissue into the space of rib segment resection on axial planes in Magnetic resonance imaging (MRI) scans performed at least 6 months postoperatively

SECONDARY OUTCOMES:
Visual contour deficit of the recipient vessels area | October 2021 to June 2023
  Postoperative photographic images were examined by two investigators (blinded to group assignments) for IMVES-associated deformities using standardized photographic images of the reconstructed breasts at the 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Dornseifer, MD/PhD, Study Director — Head of Department plastic and reconstructive surgery ISAR Klinikum
Locations (2):
- Germany (2):
  - ISAR Klinikum - Department Plastic Surgery, Munich, Bavaria
  - ISAR Klinikum, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT06504173/Prot_SAP_000.pdf